ANASTOMOTIC LEAK TEST USING INDOCYANINE

GREEN DURING LAPAROSCOPIC ROUX-EN-Y GASTRIC

**BYPASS** 

RUNNING HEADS: Indocyanine green test for evaluation of perfusion of gastro-

jejunal anastomosis during laparoscopic Roux-en-Y Gastric Bypass

NCT Number: not available

Date of document: 20/07/2022

ABSTRACT

BACKGROUND: Indocyanine green (ICG) can be injected into the human bloodstream

and it allows us to show stomach vascularity in real time. The aim of our study is to observe

the preliminary results of the application of indocyanine green fluorescence (IGF) during

laparoscopic Roux-en-Y Gastric Bypass (RYGB in our center and how the perfusion of

the gastro-jejunal anastomosis affects the onset of fistula.

MATERIALS AND METHODS: 30 consecutive patients underwent RYGB with ICG

fluorescence angiography at our center from January 2020 to December 2021. 5 ml of

ICG were then injected intravenously to identify the blood supply of the stomach and the

gastro-jejunal anastomosis.

1

RESULTS: In the RYGB tested with ICG, we all have adequate perfusion but despite this a methylene blue test was positive and allowed us to reinforce the suture of the gastrojejunal anastomosis.

CONCLUSION: Intraoperative ICG testing during laparoscopic RYGB may be helpful in determining which patients are at an increased risk for leakage but multiple factors concur to the pathophysiology and the incidence of gastric fistula not only the perfusion.

Key words: laparoscopic Roux-en-Y gastric bypass, Indocyanine green test, anastomotic fistula, gastro-jejunal leak.

#### INTRODUCTION

Morbid obesity has become a major global health threat that leads to severe morbidity including diabetes, hypertension, obstructive sleep apnea, degenerative joint dis- ease and cardiovascular diseases [1].

Bariatric surgery is recognized as the most effective treatment for morbid obesity, maintaining a stable weight reduction in the long term and reducing comorbidities, with a favorable impact on mortality [2-4].

Gastric Bypass is a common operation for weight loss in patients with severe obesity. The procedure was developed in the 1960s by Drs. Mason and Ito who observed significant weight loss in a patient undergoing partial gastrectomy for peptic ulcer disease.

As expected, any increase in the frequency of a procedure usually unveils a significant number of related complications. Most of the complications of bariatric surgery are usually observed in the postoperative period.

Ninety-day mortality is very low (less than 0.5%). The morbidity of the procedure is classified into early complications and late complications. [5]

Early complications (0-30 days):

- Venous thromboembolism (VTE)
- Anastomotic leak
- Infection
- Intestinal blockage
- Stenosis Gastro-Jejunal

# Late complications

- Intestinal blockage
- Dumping syndrome
- Marginal ulcer
- Gastrointestinal fistula
- Gallstones
- Incisional hernia
- Nutritional deficiencies

More information on complications after gastrectomy is beyond the scope of this review article. These are very complex pathological processes with specific etiologies, pathophysiology and treatments.

Gastric fistulas are the most common complication observed after gastric sleeve surgery. A meta-analysis of almost 10,000 sleeve gastrectomies conducted by Parikh et al. revealed that 2.2% of these procedures were posteriorly complicated by fistula development. In regards to Roux-en-Y gastric bypass (RYGB), anastomotic leaks are their most common complications with an incidence of 0-8% [6,7].

Indocyanine green fluorescence angiography (AF) (ICG) is an emerging technology that has been used in an attempt to reduce the incidence of anastomotic leaks. ICG is a water-

soluble tricarbocyanine dye that remains in the intravascular compartment until excretion and has a plasma half-life of between 3 and 5 minutes [8]. Importantly, the ICG absorbs light at a wavelength of excitation between 750 and 800 nm while emitting light at emission wavelengths greater than 830 nm or more [9]. Using near-infrared imaging systems, vascular perfusion to the gastro-jejunal anastomosis can be assessed intraoperatively, allowing surgeons to anastomose a well perfused bowel or to reshape a poorly perfused anastomosis. 5 ml of ICG were then injected intravenously to identify the blood supply of the stomach and the gastro-jejunal anastomosis.

The aim of our study is to observe the preliminary results of the application of indocyanine green fluorescence (IGF) during laparoscopic Roux-en-Y Gastric Bypass (RYGB in our center and how the perfusion of the gastro-jejunal anastomosis affects the onset of fistula.

#### MATERIALS AND METHODS

30 consecutive patients underwent RYGB with ICG fluorescence angiography at our center from January 2020 to December 2021.

During the period of interest, 10 male and 20 female patients underwent RYGB by the same surgical team with the same standardized technique.

The mean age was 43.6 in the male group and 37.6 in the female group (mean 39.18).

The mean preoperative BMI was roughly the same in the two groups (45.16 in the male group vs 45.06) (in the female group).

At least one major comorbidity was found in all patients: the most represented was hypertension (19 patients, 63.33%), followed by diabetes (6 patients, 20%), COPD and / or OSAS (4 patients, 12, 3%) and osteoarthritis (1 patient, 3.33%).

Five patients had previous sleeve gastrectomy surgeries.

Adequate perfusion was defined as "the direct and clear visualization of the fluorescence along the gastric tube, relative to the excised specimen, after an estimated time of 150-180 s after i.v. administration injection "(FIGURE 1a-1b).

In case of inadequate perfusion, our expected options were binding reinforcement with fibrin glue or with sutures. A methylene blue test is routinely performed after fluorescence.

The procedure ended with the placement of an intra-abdominal drain along the suture line.

On the second postoperative day, a routine swallow test with Gastrografin is performed.

After the Gastrografin swallow test, if negative, patients were given a liquid diet for 1 day, then a semi-liquid diet and were discharged on the third postoperative day.

Our follow-up was performed routinely with blood tests and clinical examination at 3-6-12 months.

Figure 1a: Evaluation of perfusion of gastro-jejunal by using Indocyanine green test

Figure 1b: Intraoperative picture of the gastro-jejunal

#### **RESULTS**

The procedure was performed in all patients without ICG-related adverse events.

Blood supply was rated "satisfactory and adequate" in all patients.

The mean operative time was 123 min. No conversion to laparotomy was performed.

Despite this, the methylene blue test was positive in only one patient, a suture reinforcement of the gastro-jejunal anastomosis was performed with Vycril stitches.

Routine swallowing of Gastrografin on the second postoperative day was negative for leaks in all patients.

No patient showed signs or symptoms of leaks at the gastro-jejunal anastomosis.

Analyzing our database, we performed 26 RYGBs without ICG tests from 2017 to 2019; the total number of leakage was 0 and our leakage rate was 0%.

In the RYGB tested with ICG, we all have adequate perfusion but despite this a methylene blue test was positive and allowed us to reinforce the suture of the gastro-jejunal anastomosis.

Furthermore, our main objective was to evaluate whether this method could adequately estimate the ischemia of the gastro-jejunal anastomosis and help in the prevention of leakage: this is so far not confirmed by our preliminary results (the only case with methylene blue test positive was adequately perfused with the ICG test).

#### **DISCUSSION**

Anastomotic leaks following RYGB can be caused by a number of factors including those compromising healing such as mechanical tension and ischemia [10] but are also associated with other factors such as BMI, age and the postoperative course [11].

The reported incidence of gastro-jejunal leakages after LRYGB has been reported to range between 1 and 3% [12-13].

The diagnosis of gastrointestinal leak after bariatric surgery can be challenging. The patient's presentation varies according to the type and timing of the leak and the patient's systemic inflammatory response. Patients with morbid obesity may show uncertain presentations, leading to late diagnosis and potentially catastrophic consequences.

There is still uncertainty about the pathophysiology of anastomotic leak after RYGB: the cause may vary from person to person. It may be caused by a problem with the tool or materials used to close the anastomosis during surgery. It may be because of problems with the blood flow in the area after surgery. Or it may be linked to other reasons for poor wound healing, such as diabetes or smoking [14-17].

The use of routine intraoperative methylene blue leak testing is still discussed as it may be useful for identifying suture line rupture but not for identifying areas at increased risk of subsequent leakage [18-20].

Recently, much interest has been focused on the possibility of assessing blood supply during surgery with the use of ICG fluorescence angiography, which is a real-time, inexpensive and feasible method of establishing vascularity in an area. [21-24]. It has been fully and positively approved in most laparoscopic procedures [25-27] but there is still little literature on its usefulness in the bariatric procedure.

Therefore, our aim was to evaluate whether intraoperative ICG fluorescence angiography could lead to estimating the ischemic area [28].

From the first data, we did not find any ischemic segmental area at the gastro-jejunal anastomosis, despite a patient with a positive methylene blue test [29-30].

### **CONCLUSIONS**

Although all patients underwent to the ICG test during RYGB showed optimal perfusion, one patient was positive to the intraoperative methylene blue test and this allowed us to reinforce the anastomosis with sutures. This information has led us to believe that multiple factors contribute to the pathophysiology and incidence of gastric fistula in the context of the RYGB operation. Therefore, intraoperative ICG testing may be helpful in determining which patients are at an increased risk for leakage, and if adjunctive measure is needed intraoperatively, but further testing is needed to determine if ICG will predict leakage due to ischemia.

## REFERENCES

- 1. Younis F, Shnell M, Gluck N, Abu-Abeid S, Eldar S, Fishman S. Endoscopic treatment of early leaks and strictures after laparoscopic one anastomosis gastric bypass. BMC Surg. 2020 Feb 21;20(1):33. doi: 10.1186/s12893-020-0686-2. PMID: 32085769; PMCID: PMC7035723.
- 2. Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, et al. Bariatric surgery:a systematic review and meta-analysis. JAMA. 2004;292(14):1724-37.
- 3. Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, et al. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004;240(3):416-23; discussion 423-4.
- 4. Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, et al. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007;357(8):741-52.

- Peterli R, Wölnerhanssen BK, Peters T, Vetter D, Kröll D, Borbély Y, Schultes B, Beglinger C, Drewe J, Schiesser M, Nett P, Bueter M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss in Patients With Morbid Obesity: The SM-BOSS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):255-265. doi: 10.1001/jama.2017.20897. PMID: 29340679; PMCID: PMC5833546.
- 6. Surgical strategies that may decrease leak after laparoscopic sleeve gastrectomy: a systematic review and meta-analysis of 9991 cases. Parikh M, Issa R, McCrillis A, Saunders JK, Ude-Welcome A, Gagner M. *Ann Surg.* 2013;257:231–237. [PubMed] [Google Scholar]
- 7. Diagnosis and management of the postoperative surgical and medical complications of bariatric surgery. Montravers P, Augustin P, Zappella N, et al. *Anaesth Crit Care Pain Med.* 2015;34:45–52. [PubMed] [Google Scholar]
- 8. Keller DS, Ishizawa T, Cohen R, Chand M. Indocyanine green fluorescence imaging in colorectal surgery: overview, applications, and future directions. Lancet Gastroenterol Hepatol. 2017;2:757e766.
- 9. Alander JT, Kaartinen I, Laakso A, et al. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585.
- 10. Gonzalez R, Nelson LG, Gallagher SF, et al. Anastomotic leaks after laparoscopic gastric bypass. *Obes Surg.* 2004;14:1299–307.
- 11. Ballesta C, Berindoague R, Cabrera M, et al. Management of anastomotic leaks after laparoscopic Roux-en-Y gastric bypass. *Obes Surg.* 2008;18:623–30.
- 12. Singhal R, Tahrani AA, Ludwig C, Mahawar K; GENEVA collaborators. Global 30-day outcomes after bariatric surgery during the COVID-19 pandemic (GENEVA): an international cohort study. Lancet Diabetes Endocrinol. 2021 Jan;9(1):7-9. doi: 10.1016/S2213-8587(20)30375-2. Epub 2020 Nov 27. PMID: 33253631; PMCID: PMC7832244.
- 13. Flum DR, Belle SH, King WC, et al: Periop- erative safety in the longitudinal assessment of bariatric surgery. N Engl J Med 2009;361: 445–454.

- 14. Alizadeh RF, Li S, Inaba C, Penalosa P, Hinojosa MW, Smith BR, Stamos MJ, Nguyen NT. Risk Factors for Gastrointestinal Leak after Bariatric Surgery: MBASQIP Analysis. J Am Coll Surg. 2018 Jul;227(1):135-141. doi: 10.1016/j.jamcollsurg.2018.03.030. Epub 2018 Mar 30. PMID: 29605723.
- 15. Tartaglia N, Pavone G, Di Lascia A, Vovola F, Maddalena F, Fersini A, Pacilli M, Ambrosi A. Robotic voluminous paraesophageal hernia repair: a case report and review of the literature. J Med Case Rep. 2020 Feb 4;14(1):25. doi: 10.1186/s13256-020-2347-6. PMID: 32019608; PMCID: PMC6998085.
- 16. Pacilli M, Tartaglia N, Gerundo A, Pavone G, Fersini A, Ambrosi A. Energy Based Vessel Sealing Devices in Thyroid Surgery: A Systematic Review to Clarify the Relationship with Recurrent Laryngeal Nerve Injuries. Medicina (Kaunas). 2020 Nov 27;56(12):651. doi: 10.3390/medicina56120651. PMID: 33260912; PMCID: PMC7760641
- 17. Tartaglia N., Pavone G., Petruzzelli F., Di Lascia A., Vovola F., Maddalena F., Cianci P., Fersini A., Pacilli M., Ambrosi A. Robotic sleeve gastrectomy vs laparoscopic sleeve gastrectomy: our preliminary experience and a literature review. Clinical and Experimental Surgery. Petrovsky Journal. 2020; 8 (4): 7–15. DOI: https://doi.org/10.33029/2308-1198-2020-8-4-7-15
- 18. Singhal R, Ludwig C, Rudge G, Gkoutos GV, Tahrani A, Mahawar K; GENEVA Collaborators, et al. 30-Day Morbidity and Mortality of Bariatric Surgery During the COVID-19 Pandemic: a Multinational Cohort Study of 7704 Patients from 42 Countries. Obes Surg. 2021 Oct;31(10):4272-4288. doi: 10.1007/s11695-021-05493-9. Epub 2021 Jul 30. PMID: 34328624; PMCID: PMC8323543.
- 19. Tartaglia N, Pavone G, Lizzi V, Vovola F, Tricarico F, Pacilli M, Ambrosi A. How emergency surgery has changed during the COVID-19 pandemic: A cohort study. Ann Med Surg (Lond). 2020 Dec 5;60:686-689. doi: 10.1016/j.amsu.2020.12.001. PMID: 33312562; PMCID: PMC7719013.
- 20. Benedix F, Benedix DD, Knoll C et al. Are there risk factors that in- crease the rate of staple line leakage in patients undergoing primary sleeve gastrectomy for morbid obesity? ObesSurg 2014; 24: 1610–1616

- 21. Sakran N, Goitein D, Raziel A, et al. Gastric leaks after sleeve gastrectomy: a multicenter experience with 2,834 patients. SurgEndosc. 2013;27(1):240–5. https://doi.org/10.1007/s00464-012- 2426-x
- 22. Benedix F, Benedix DD, Knoll C, et al. Are there risk factors that increase the rate of staple line leakage in patients undergoing pri- mary sleeve gastrectomy for morbid obesity? ObesSurg. 2014;24(10):1610–6.
- 23. Lacedonia D, Tartaglia N, Scioscia G, Soccio P, Pavone G, Moriondo G, Gallo C, Foschino Barbaro MP, Ambrosi A. Different Expression of Micro-RNA in the Subcutaneous and Visceral Adipose Tissue of Obese Subjects. Rejuvenation Res. 2022 Apr;25(2):89-94. doi: 10.1089/rej.2022.0004. PMID: 35293246.
- 24. Singhal R, Cardoso VR, Wiggins T, Super J, Ludwig C, Gkoutos GV, Mahawar K; GENEVA Collaborators. 30-day morbidity and mortality of sleeve gastrectomy, Roux-en-Y gastric bypass and one anastomosis gastric bypass: a propensity score-matched analysis of the GENEVA data. Int J Obes (Lond). 2022 Apr;46(4):750-757. doi: 10.1038/s41366-021-01048-1. Epub 2021 Dec 15. PMID: 34912046; PMCID: PMC8671878.
- 25. Delle Monache S, Calgani A, Sanità P, et al. Adipose-derived stem cells sustain prolonged angiogenesis through leptin secretion. GrowthFactors. 2016;34(3–4):87–96. https://doi.org/10.1080/08977194.2016.1191481.
- 26. Cobianchi L, Dal Mas F, Massaro M, Fugazzola P, Coccolini F, Kluger Y, Leppäniemi A, Moore EE, Sartelli M, Angelos P, Catena F, Ansaloni L; Team Dynamics Study Group. Team dynamics in emergency surgery teams: results from a first international survey. World J Emerg Surg. 2021 Sep 16;16(1):47. doi: 10.1186/s13017-021-00389-6. Erratum in: World J Emerg Surg. 2021 Nov 1;16(1):55. PMID: 34530891; PMCID: PMC8443910.
- 27. Tartaglia N, Di Lascia A, Cianci P, Fersini A, Pacilli M, Pavone G, Ambrosi A. Hemoperitoneum caused by spontaneous rupture of hepatocellular carcinoma in noncirrhotic liver. A case report and systematic review. Open Med (Wars). 2020 Aug 3;15(1):739-744. doi: 10.1515/med-2020-0202. PMID: 33336031; PMCID: PMC7712383.

- 28. Singhal R, Wiggins T, Super J, Alqahtani A, Nadler EP, Ludwig C, Tahrani A, Mahawar K; GENEVA Collaborative. 30-Day morbidity and mortality of bariatric metabolic surgery in adolescence during the COVID-19 pandemic The GENEVA study. Pediatr Obes. 2021 Dec;16(12):e12832. doi: 10.1111/ijpo.12832. Epub 2021 Jul 8. PMID: 34240553.
- 29. Cianci P, Tartaglia N, Altamura A, Di Lascia A, Fersini A, Neri V, Ambrosi A. Cervical Esophagotomy for Foreign Body Extraction: A Case Report and Extensive Literature Review of the Last 20 Years. Am J Case Rep. 2018 Apr 5;19:400-405. doi: 10.12659/ajcr.908373. PMID: 29618719; PMCID: PMC5900799.
- 30. Tartaglia N, Iadarola R, Di Lascia A, Cianci P, Fersini A, Ambrosi A. What is the treatment of tracheal lesions associated with traditional thyroidectomy? Case report and systematic review. World J Emerg Surg. 2018 Mar 23;13:15. doi: 10.1186/s13017-018-0175-4. PMID: 29588652; PMCID: PMC5865337.

Provenance and peer review

Not commissioned, externally peer-reviewed